CLINICAL TRIAL: NCT03058913
Title: OEIS (Outpatient Endovascular and Interventional Society) Outcome Data Registry
Brief Title: OEIS Outcome Data Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Outpatient Endovascular and Interventional Society (Other)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Other Study IDs: 2016-OEIS-01
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry is created under the sponsorship of the Outpatient Endovascular and Interventional Society (OEIS) to monitor the clinical course and treatment outcomes of patients undergoing office-based endovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older;
* Patient is identified as having undergone a percutaneous transluminal vascular intervention or attempted intervention, in an ambulatory (outpatient) facility, for the treatment of peripheral vascular disease within native arteries or bypass grafts, from the infrarenal aorta distally to the feet.

Exclusion Criteria:

* Patient treated for a non-eligible condition or procedure
* Diagnostic procedures without intervention or attempted interventions
* Serious mental illness that might preclude subject's ability to comply with follow up
* Life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the registry diagnostic and procedure inclusion criteria and that are treated at participating facilities by participating clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 600000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Antiplatelet Therapy (ACC/AHA/PAD Coalition) | 30 days
  To collect the clinical variables of Patients undergoing endovascular procedures in an outpatient angiograPercentage of patients with PAD that have been prescribed an antiplatelet medication at the reported encounter.
Preventive Care and Screening: Tobacco Use | 30 days
  Screening and Cessation Intervention. Percentage of patients aged 18 years and older who were screened for tobacco use one or more times within 24 months AND who received cessation counseling intervention if identified as a tobacco user.
Lipid-Lowering Medications for Patients with PAD | 30 days
  The rate at which patients with documented peripheral artery disease have documentation of a currently prescribed antihyperlipidemic medication treatment. This may include one of the following: Statin, Bile acid sequestrants, Niacin, Ezetemibe, Fibrates, PCSK9 Inhibitors
Optimal vascular care | 30 days
  This measure is a composite score of appropriate vascular care measures for treatment of PAD. This measure is a composite result of 1: Antiplatelet Therapy; 2: Preventive Care and Screening: Tobacco Use; and 3: Lipid-Lowering Medications (Statin) for Patients with PAD
Preventive Care and Screening: Influenza Immunization. | 30 days
Pneumonia Vaccination Status for Older Adults. | 30 days
Preventive Care and Screening: Screening for High Blood Pressure and Follow-Up Documented. | 30 days
Appropriate non-invasive arterial testing for patients with intermittent claudication who are undergoing a lower extremity peripheral vascular intervention. | 30 days
  Proportion of patients with non-invasive evaluations present/available prior to lower extremity peripheral vascular interventions in patients with intermittent claudication.
Appropriate non-invasive arterial testing for patients with critical limb ischemia who are undergoing a LE peripheral vascular intervention. | 30 days
  Proportion of patients with non-invasive evaluations present/available prior to LE peripheral vascular interventions in patients with critical limb ischemia.
Emergent transfer from an outpatient, ambulatory surgical center, or office setting. | 30 days
  Rate of emergent transfer from an outpatient, ASC, or office setting to an acute care facility as a result of an invasive peripheral vascular intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Endovascular Interventional Society (OEIS), Hoffman Estates, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carey K, Burgess JF Jr, Young GJ. Hospital competition and financial performance: the effects of ambulatory surgery centers. Health Econ. 2011 May;20(5):571-81. doi: 10.1002/hec.1617. PMID 21433218
- [Background] Murer CG. Significant changes for ASC payment systems. Rehab Manag. 2007 Nov;20(9):42, 44-5. No abstract available. PMID 18229814
- [Background] Lapetina EM, Armstrong EM. Preventing errors in the outpatient setting: a tale of three states. Health Aff (Millwood). 2002 Jul-Aug;21(4):26-39. doi: 10.1377/hlthaff.21.4.26. PMID 12117139
- [Background] Kutscher B. Outpatient care takes the inside track. Mod Healthc. 2012 Aug 6;42(32):24-6. No abstract available. PMID 22953497
- [Background] Lin PH, Yang KH, Kollmeyer KR, Uceda PV, Ferrara CA, Feldtman RW, Caruso J, Mcquade K, Richmond JL, Kliner CE, Egan KE, Kim W, Saines M, Leichter R, Ahn SS. Treatment outcomes and lessons learned from 5134 cases of outpatient office-based endovascular procedures in a vascular surgical practice. Vascular. 2017 Apr;25(2):115-122. doi: 10.1177/1708538116657506. Epub 2016 Jul 9. PMID 27381926